CLINICAL TRIAL: NCT01848860
Title: Thoracoscopic Bullectomy With Absorbable Mesh Coverage of the Staple Line Versus Thoracoscopic Bullectomy Only for the Treatment of Primary Spontaneous Pneumothorax: a Single-blind, Parallel-group, Prospective, Randomized Controlled Trial
Brief Title: Absorbable Mesh Pleurodesis in Thoracoscopic Treatment of Spontaneous Pneumothorax
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201211051DIC
Record Dates: First submitted 2013-05-04; First posted 2013-05-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Spontaneous Pneumothorax; Surgery
Keywords: Pneumothorax; thoracoscopy; mesh; pleurodesis; treatment
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Sham Comparator): In this group, only thoracoscopic bullectomy and pleural abrasion will be done.
  Interventions: Procedure: Thoracoscopic bullectomy and pleural abrasion
- Mesh group (Experimental): In this group, absorbable mesh coverage of the staple line will be performed after thoracoscopic bullectomy and pleural abrasion.
  Interventions: Procedure: Thoracoscopic bullectomy and pleural abrasion; Biological: Mesh coverage of the staple line

INTERVENTIONS:
Procedure: Thoracoscopic bullectomy and pleural abrasion — Thoracoscopic bullectomy and pleural abrasion will be performed in a standard fashion under general anesthesia using intubated one-lung ventilation. When blebs are identified, they will be grasped with the ring forceps and excised with an endoscopic stapler. Blind apical stapling was done at the most suspicious area if no bleb could be identified. Thoracoscopic pleural abrasion will be performed at the parietal pleura above the 5th intercostal space by inserting the dissector with a strip of diathermy scratch pad through the port sites in all patients.
Biological: Mesh coverage of the staple line — Absorbable mesh coverage of the staple line will be performed in the mesh group after thoracoscopic bullectomy in the mesh group
  Arms: Mesh group

SUMMARY:
Primary spontaneous pneumothorax usually occurs in young, lean male without underlying lung disease. In most cases, the cause of pneumothorax is rupture of blebs at the apex of the lung. Traditionally, bullectomy with mechanical pleurodesis through thoracotomy is indicated in patients with recurrence or persisted air leakage. In recent years, thoracoscopic bullectomy with pleural abrasion is getting popular, thanks for the advance of endoscopic instruments and technique. The pneumothorax recurrence rate after thoracoscopic surgery is around 10%, which is significantly higher than that of thoracotomy. In addition, the rate of postoperative prolonged air leakage is 5-8%. The possible causes of recurrent pneumothorax and prolonged air leakage are missed bleb surrounding the endoscopic suture line or suboptimal suturing or healing of the thoracoscopic suture. To prevent these complications, a novel method using coverage of the endoscopic suture line by a large absorbable mesh during thoracoscopic surgery was proved to be safe and feasible. Theoretically, the mesh can strengthen the suture line and induce local fibrosis surrounding the suture line, and reduce the rate of recurrent pneumothorax and prolonged air leakage. To prove this hypothesis, the investigators are conducting a prospective randomized trial in National Taiwan University Hospital. The investigators will enroll 204 patients with primary spontaneous pneumothorax who will be randomly assigned to additional mesh pleurodesis (mesh group, 102 patients) or not (control group, 102 patients) after thoracoscopic bullectomy and pleural abrasion. The primary endpoint is to compare the rate of pneumothorax recurrence within one year between the two groups. The secondary endpoints are to compare the safety, efficacy, and long-term pulmonary function between the two groups.

DETAILED DESCRIPTION:
Primary spontaneous pneumothorax most commonly occurs in young, tall, lean males (1, 2). The estimated recurrence rate is 23-50% after the first episode and increases to 60% after the second pneumothorax (3). Optimal management of this benign disease, especially after repeat attack, has been a matter of debate. Recent advances in video-assisted thoracoscopic surgery (VATS) that combine bullectomy with pleural abrasion provide a preferred intervention for treating primary spontaneous pneumothorax (4-6). Unfortunately, recurrence rates of pneumothorax after VATS range between 5% and 10%, which are higher than the rates reported after open thoracotomy (7-11). It is suggested that a higher chance of missed leaking blebs around the staple line of endoscopic staplers (12) and a less intense pleural inflammatory reaction are induced by VATS procedure than by thoracotomy (13, 14). In addition, postoperative air leakage usually occurs at the staple line. (7, 15) As a result, the efficacy of VATS is questioned and more aggressive procedures, such as limited thoracotomy with pleurectomy, are sometimes performed to enhance the effects of pleural symphysis (10, 14).

Theoretically, reinforcement of the visceral pleura around the staple line is a reasonable way to prevent postoperative air leak and recurrent pneumothorax. Previous retrospective studies showed that staple line coverage with absorbable mesh after thoracoscopic bullectomy is safe and may be effective in decreasing the rates of pneumothorax recurrence (16,17). One animal study also showed that when absorbable mesh insertion is coupled with pleural abrasion, appropriate pleurodesis is predictably achieved (18).

In the present study, additional absorbable mesh coverage of the staple line will be randomly administered in patients with primary spontaneous pneumothorax after VATS to test the efficacy and safety of this method.

References

1. Gobbel WG Jr, Rhea WG, Nelson IA, Daniel RA Jr. Spontaneous pneumothorax. J Thorac Cardiovasc Surg 1963;46:331-345.
2. Lichter J, Gwynne JF. Spontaneous pneumothorax in young subjects. Thorax 1971;25:409-417.
3. Light RW. Management of spontaneous pneumothorax. Am Rev Respir Dis 1993;148:245-258.
4. Baumann MH, Strange C, Heffner JE, Light R, Kirby TJ, Klein J, Luketich JD, Panacek EA, Sahn SA; AACP Pneumothorax Consensus Group. Management of spontaneous pneumothorax: an American College of Chest Physicians Delphi consensus statement. Chest 2001;119:590-602.
5. Naunheim KS, Mack MJ, Hazelrigg SR, Ferguson MK, Ferson PF, Boley TM, Landreneau RJ. Safety and efficacy of video-assisted thoracic surgical techniques for the treatment of spontaneous pneumothorax. J Thorax Cardiovasc Surg 1995;109:1198-1204.
6. Mouroux J, Elkaim D, Padovani B, Myx A, Perrin C, Rotomondo C, Chavaillon JM, Blaive B, Richelme H. Video-assisted thoracoscopic treatment of spontaneous pneumothorax: technique and results of one hundred cases. J Thorac Cardiovasc Surg 1996;112:385-391.
7. Hatz RA, Kaps MF, Meimarakis G, Loehe F, Muller C, Furst H. Long-term results after video-assisted thoracoscopic surgery for first-time and recurrent spontaneous pneumothorax. Ann Thorac Surg 2000;70:253-257.
8. Inderbitzi RG, Leiser A, Furrer M, Althaus U. Three years' experience in video-assisted thoracic surgery (VATS) for spontaneous pneumothorax. J Thorac Cardiovasc Surg 1994;107:1410-1415.
9. Chan P, Clarke P, Daniel FJ, Knight SR, Seevanayagam S. Efficacy study of video-assisted thoracoscopic surgery pleurodesis for spontaneous pneumothorax. Ann Thorac Surg 2001;71:452-454.
10. Massard G, Thomas P, Wihlm JM. Minimally invasive management for first and recurrent pneumothorax. Ann Thorac Surg 1998;66:592-599.
11. Sahn SA, Heffner JE. Spontaneous pneumothorax. N Engl J Med 2000;342:868-874.
12. Sakamoto K, Kase M, Mo M, et al. Regrowth of bullae around the staple-line is one of the causes of postoperative recurrence in thoracoscopic surgery for spontaneous pneumothorax. Kyobu Geka 1999;52:939-42.
13. Gebhard FT, Becker HP, Gerngross H, Bruckner UB. Reduced inflammatory response in minimally invasive surgery of pneumothorax. Arch Surg 1996;131:1079-1082.
14. Horio H, Nomori H, Fuyuno G, Naruke T, Suemasu K. Limited axillary thoracotomy vs video-assisted thoracoscopic surgery for spontaneous pneumothorax. Surg Endosc 1998:12:1155-1158.
15. How CH, Tsai TM, Duo SW, et al. Chemical pleurodesis for prolonged postoperative air leak in primary spontaneous pneumothorax. J Formos Med Assoc, accepted.
16. Nakanishi K. An apical symphysial technique using a wide absorbable mesh placed on the apes for primary spontaneous pneumothorax. Surg Endosc 2009;23:2515-2521.
17. Sakamoto K, Takei H, Nishii T, et al. Staple line coverage with absorbable mesh after thoracoscopic bullectomy for spontaneous pneumothorax. Surg Endosc 2004;18:478-481.
18. Suqarmann WM, Widmann WD, Mysh D, et al. Mesh insertion as an aid for pleurodesis. J Cardiovasc Surg 1996;37:173-5.

ELIGIBILITY:
Inclusion criteria:

1. Age between 15 and 50 years old.
2. Spontaneous pneumothorax requiring thoracoscopic surgery.
3. With written inform consent

Exclusion criteria:

1. With underlying pulmonary disease (chronic obstructive pulmonary disease, bronchiectasis, tuberculosis, etc)
2. A history of previous ipsilateral thoracic operation
3. Diagnosis of catamenial pneumothorax
4. Diagnosis of lymphangioleiomyomatosis
5. Concurrent hemopneumothorax with bleeding > 500ml/h
6. Pregnant or lactating women
7. Other serious concomitant illness or medical conditions:

   1. Congestive heart failure or unstable angina pectoris.
   2. History of myocardial infarction within 1 year prior to the study entry.
   3. Uncontrolled hypertension or arrhythmia.
   4. History of significant neurologic or psychiatric disorders, including dementia or seizure.
   5. Active infection requiring i.v. antibiotics.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 204 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the rates of ipsilateral pneumothorax recurrence | 12 months
  The detection of pneumothorax recurrence will be performed by chest radiography

SECONDARY OUTCOMES:
Safety of mesh coverage | 30 days
  Early postoperative results, including postoperative pain scores, postoperative duration of chest drainage, postoperative duration of hospital stay, and complication rates.
long-term safety of mesh coverage | 12 months
  Long-term results, including residual chest pain at 6 months, and postoperative pulmonary function at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Hsu HH, Liu YH, Chen HY, Chen PH, Chen KC, Hsieh MJ, Lin MW, Kuo SW, Huang PM, Chao YK, Wu CF, Wu CY, Chiu CH, Chen WH, Wen CT, Liu CY, Wu YC, Chen JS. Vicryl Mesh Coverage Reduced Recurrence After Bullectomy for Primary Spontaneous Pneumothorax. Ann Thorac Surg. 2021 Nov;112(5):1609-1615. doi: 10.1016/j.athoracsur.2020.11.012. Epub 2021 May 1. PMID 33279544